CLINICAL TRIAL: NCT03607695
Title: Genetic Influences on Response to Gait Rehabilitation in Parkinson's Disease
Acronym: Gen-Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: E2553-P; I21RX002553-01 (NIH)
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Parkinson's Disease
Keywords: gait; exercise; cognition; genetics
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: The intervention is a 10-week gait, treadmill-training program. The sessions are 1 hour long, twice a week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gait training (Experimental): 1 hour walking exercise on a treadmill
  Interventions: Other: Gait training

INTERVENTIONS:
Other: Gait training — Walking on a treadmill and receiving audio cues to improve gait

SUMMARY:
The aging Veteran population, together with high exposure to Agent Orange or other herbicides during military service, has made diseases such as Parkinson's disease (PD), currently affecting more than 80,000 Veterans, a major health issue in the Veterans' health system. Mobility and cognitive limitations are a common problem in PD and are associated with significant disability, increased fall risk, reduced quality of life, and increased caregiver burden. While less is known about its benefit on cognition, physical therapy has proven to be an effective treatment to mitigate mobility limitations, though the response to rehabilitation interventions is highly variable. The proposed research will inform the investigators' understanding of the impact of certain genetic profiles associated with learning impairments on motor and cognitive benefits in response to gait rehabilitation, and will provide an important foundation for more personalized and improved gait rehabilitation programs for different subgroups of PD patients.

DETAILED DESCRIPTION:
The completion of the Human Genome Project in 2003 marked the beginning of the genomic era and the birth of "personalized" (precision) medicine. In the last decade, genetics have provided a new understanding of predicting, diagnosing, and treating individual health conditions. Indeed, such precision medicine has begun to impact virtually all areas of medicine, with significant potential to influence the timing, dosage, and intensity of physical rehabilitation.

The long-term goals of this research are: (1) to determine if certain genetic variants associated to learning impairments impact the motor and cognitive benefit experienced in response to physical rehabilitation in Veterans with Parkinson's disease (PD), and (2) to use that knowledge to identify subpopulations of patients that may require rehabilitative strategies tailored to their genotype to optimize physical rehabilitation. To achieve these goals the investigators will enroll 30 Veterans with PD in a 10-week moderate intensity gait training program consisting of 2 times per week treadmill training with verbal cues for gait quality. Aim 1 will examine the association between variants in 2 genes known to affect cognition and motor learning (APOE- 4 and BDNF-Met66), and motor improvements after gait training. Specifically, changes in walking from during and after training will be sensitively and objectively assessed using state-of-the-art quantitative gait analysis, and compared between three genotype groups (carriers of BDNF-Met66 (N=10), carriers of APOE- 4 (N=10) and those not carrying either of those variants (N=10)). Aim 2 will examine the effect of APOE- 4 and BDNF-Met66 genetic variants on cognitive changes in response to this training program. In order to do this the investigators will measure cognitive performance pre- and post-training using a brief, targeted battery aimed at assessing attention, processing speed, executive function, and learning/memory, the domains more affected, and more likely to improve with physical exercise in PD. The investigators will test the hypothesis that Veterans with PD who carry an APOE- 4 or BDNF-Met66 allele will demonstrate smaller improvements in gait (Aim 1) and cognition (Aim 2) in response to a 10-week gait training program. Overall the results of this project will enhance the investigators' knowledge regarding the influence of different genetic profiles in the response to physical rehabilitation in Veterans with PD, and will generate supporting data that will translate to more personalized and effective rehabilitation programs for people with PD.

ELIGIBILITY:
Inclusion Criteria:

* Meet UK Brain Bank (UKBB) criteria for the diagnosis of PD (modified so that having more than one affected relative was not considered an exclusion criteria)
* Have a Hoehn & Yahr score of 3
* Have the ability to walk 400 m without physical assistance from a device or another person
* Do not have other health conditions (e.g., orthopedic, cardiopulmonary) that impact the ability to safely participate in a moderately intense gait training program

Exclusion Criteria:

* The investigators will exclude those patients presenting clinical diagnosis of dementia.
* The investigators will exclude those patients presenting conditions (cardiac, renal, or metabolic) that would pose a risk to their health by exercising.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Fernandez-Mata, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
We will not make individual participant data available.

RESULTS

PARTICIPANT FLOW:
Groups:
- Gait Training: 1 hour walking exercise on a treadmill
  Gait training: Walking on a treadmill and receiving verbal cues to improve gait quality
Period: 2 Week
Arm/Group | Gait Training
Started | 19
Completed | 19
Not Completed | 0
Period: 10 Week
Arm/Group | Gait Training
Started | 19
Completed | 18
Not Completed | 1
Not completed — Local and institutional restrictions on research enacted due to COVID-19 pandemic | 1
Period: 16 Week
Arm/Group | Gait Training
Started | 18
Completed | 16
Not Completed | 2
Not completed — Local and institutional restrictions on research enacted due to COVID-19 pandemic | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gait Training
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Gait Speed (m/s)
Description: The investigators will use the APDM Movement Monitoring system to assess gait speed (m/s) during straight-line walking as a measure of gait function.
Time Frame: measured at baseline, 2 weeks, 10 weeks and 16 weeks
Population: Three participants did not complete the 16 week (follow-up) visit due to local and institutional restrictions on research implemented early in the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Gait Training
Number analyzed (Participants) | 19
m/s
  Baseline | 1.14 (0.16)
  2 week | 1.21 (0.16)
  10 week | 1.22 (0.17)
  16 week: number analyzed (Participants) | 16
  16 week | 1.20 (0.12)

2. Primary Outcome: Montreal Cognitive Assessment Score
Description: The investigators will use the Montreal Cognitive Assessment (MoCA; score range=0-30, with 30 indicating better cognitive function) as a reflection of global cognitive function
Time Frame: measured at baseline and at 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gait Training
Number analyzed (Participants) | 19
score on a scale
  Baseline | 27.1 (1.6)
  Week 10 | 27.7 (2.0)

ADVERSE EVENTS:
Time Frame: 16 weeks (study duration)
Arm/Group | Gait Training
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 6/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gait Training (N=19)
Fall (outside of study visit) (General disorders) | 2 (2) — Fall reported outside of study visits
Lightheadedness (General disorders) | 1 (1) — Hypotensive episode after study visit
Exercise-associated pain, fatigue (Musculoskeletal and connective tissue disorders) | 3 (3) — Muscle pain, joint pain, fatigue after intervention session

LIMITATIONS AND CAVEATS:
This trial was impacted by local and institutional restrictions on research implemented during the start of the COVID-19 pandemic. Restrictions on research activities impacted recruitment and impacted data collection for some participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT03607695/Prot_SAP_000.pdf